CLINICAL TRIAL: NCT01115296
Title: Control of Helicobacter Pylori Infection by Dietary Supplementation With Lactobacillus Reuteri
Brief Title: Control of Helicobacter Pylori Infection by Probiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, MD, PhD, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-Progastria
Record Dates: First submitted 2010-04-28; First posted 2010-05-04 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter Pylori; gastritis; Probiotics; Lactobacillus Reuteri
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 'L. reuteri DSM 17938 and ATCC PTA 6475 (Active Comparator): L. reuteri will be delivered at a dose of 1x108 CFU of each strain of L. reuteri giving a final dose of L. reuteri of 2x108 CFU. One dose is to be taken once per day giving a dose of L. reuteri of 2x108 CFU/day.
  Interventions: Dietary Supplement: L. reuteri DSM 17938 and ATCC PTA 6475
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938 and ATCC PTA 6475 — L. reuteri dose of 1x108 CFU.
  Other Names: Probiotic mixture
  Arms: 'L. reuteri DSM 17938 and ATCC PTA 6475
Other: Placebo — Placebo
  Other Names: Placebo identical to active
  Arms: Placebo

SUMMARY:
Helicobacter pylori colonises an estimated 50% of the world´s population (Taylor & Blaser, 1991; Go, 2002). Despite clear clinical guidelines on the treatment of this infection (Malfertheiner et al. 2007) there is a drive to find alternative ways to control this infection in a wider perspective without the complications of induction of antibiotic resistance in the pathogen.

L. reuteri has been widely studied in clinical trials and has been shown to have probiotic, health-promoting effects in both adults and children (Connolly 2004; Casas & Dobrogosz, 2000). L. reuteri has been shown in numerous studies to be safe for human consumption and it has been shown to colonise the human gastrointestinal tract (Wolf et al., 1995, Valeur et al., 2004).

Studies using supplementation with L. reuteri in both symptomatic and non-symptomatic H. pylori-infected subjects show a clear reduction of infection load after 4 weeks of use and this was concomitant with a reduction in symptoms associated with the infection (Imase et al. 2007; Francavilla et al. 2007, unpublished data). Further, dietary supplementation with L. reuteri during and after the period of H. pylori eradication therapy has also been shown to reduce the side effects of this therapy without affecting the degree of eradication (Lionetti et al., 2007). It is also feasible, through the inhibitory action of L. reuteri on H. pylori, that pre-exposure to L. reuteri may weaken H. pylori and make it more susceptible to antibiotic attack during eradication.

However, an earlier pilot study was not been able to demonstrate a reduction in gastric inflammation caused by H. pylori. This pilot study was performed with L. reuteri ATCC 55730 that has since been found to lack anti-inflammatory activity in in vitro screens. Recent selection of natural, human L. reuteri strains has identified a specific strain with strong anti-inflammatory properties in vitro (Lin et al, 2007 and submitted 2007). A combination of this strain, together with the earlier proven L. reuteri strain, is expected to lead to both a reduction of H. pylori load as well as a reduction in the gastric inflammation related to the pathogen.

DETAILED DESCRIPTION:
INVESTIGATIONAL PLAN AND PROCEDURES Randomised, double-blind, placebo-controlled clinical trial. One hundred (100) subjects, aged 18-65 years recruited from patients with symptoms referred for consultation about H. pylori infection naive to treatment. HP infected patients will then be randomly allocated to two groups, one to receive L. reuteri and the other to receive an identical placebo preparation.

Baseline tests:

1. 13C-UBT
2. Gastrointestinal symptom rating score (GSRS)
3. Serological assessment of H. pylori
4. Measurement of marker serum peptides related to gastric inflammation.

The subjects will be asked to take the study product each day for 28 days. On Day 29, the subjects will return to the clinic for repeated analysis of:

1. 13C-UBT
2. Gastrointestinal symptom rating score (GSRS)
3. Measurement of marker serum peptides related to gastric inflammation.
4. Endoscopy with the collection of 5 gastric biopsy samples (4 from the antrum and 1 from the corpus).

After this analysis (Day 29), eradication treatment will be initiated. Patients will receive lansoprazole (30 mg b.d.) plus amoxycillin (1 gr b.d.) for 5 days followed by lansoprazole (30 mg b.d.) plus clarithromycin (250 b.d.) and tinidazole (500 b.d.) for the next 5 days, as recommended in the Maastricht III criteria (Malfertheiner et al. (2007).

The study products will be administered throughout the eradication treatment period of 10 days. At the end of eradication therapy all subjects will return to the clinic for repeated analysis of:

1. Gastrointestinal symptom rating score (GSRS)
2. Measurement of marker serum peptides related to gastric inflammation. At this visit patients will be given a GSRS questionnaire to complete at home 30 days after this visit. The completed GSRS shall be given to the investigators at the final visit by the patient.

The subjects will continue to take the study product for a further 60 days after the completion of eradication. After this further 60 days (to allow discrimination between recrudescence and re-infection), the level of eradication of H. pylori and the symptom score will again be analysed

1. 13C-UBT
2. Gastrointestinal symptom rating score (GSRS)
3. Measurement of marker serum peptides related to gastric inflammation.

Concomitant treatment During the period of the study (other than during the eradication therapy), the subjects will refrain from ingestion of any kind of probiotic or bacterial preparation, antibiotics, H2-antagonists, PPIs and NSAIDs.

Study Product and Dosage L. reuteri Progastria consists of a mixture of two human strains of L. reuteri, L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475. L. reuteri DSM 17938 is essentially the same strain as L. reuteri ATCC 55730, except that it lacks plasmids that carried antibiotic resistance traits for tetracycline and lincomycin. This strain has been extensively studied in humans of all ages. L. reuteri ATCC PTA 6475 is a new strain that was isolated from the breast milk of a nursing mother (as was L. reuteri DSM 17938).

L. reuteri will be delivered at a dose of 1x108 CFU of each strain of L. reuteri giving a final dose of L. reuteri of 2x108 CFU. One dose is to be taken once per day giving a dose of L. reuteri of 2x108 CFU/day. This dose of L. reuteri has been shown to be effective in a series of conditions earlier, including inhibition of H. pylori in humans, and is considered the optimal dose.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 - 65 years
* Infection with H. pylori defined as ∆ > 20 ppm in the UBT test
* Non-ulcer dyspepsia
* No earlier eradication therapy for H. pylori infection
* Written informed consent
* Stated availability throughout the entire study period
* Mental ability to understand and willingness to fulfil all the details of the protocol.

Exclusion Criteria:

* Duodenal or gastric ulcer
* MALT lymphoma
* Gastric resection (at any time)
* First level relatives of gastric cancer patients
* Absence of GI symptoms
* Use of NSAIDs, aspirin or other anti-inflammatory drugs within 1 week (for occasional use) or 3 weeks (for chronic use) of inclusion
* Use of oral antibiotics and/or PPIs and/or H2-antagonists during the 2 weeks prior to ingestion of the study product
* Pregnancy
* Participation in other clinical trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
to decrease H. pylori gastric load | 28 days
  Primary Outcome Measures:
  Decrease H. pylori gastric load by histology after 28 days compared to placebo and by 13C-UBT compared to placebo.

SECONDARY OUTCOMES:
To decrease dyspeptic symptoms | 28 days
  To decrease dyspeptic symptoms before, during and after eradication therapy as assessed by a gastro-intestinal symptom rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Principi Beatrice, MD, Principal Investigator — University of Bari
Locations (1):
- Unit of Gastroenterology, Bari, Italy, Italy

REFERENCES:
- [Background] Francavilla R, Lionetti E, Castellaneta SP, Magista AM, Maurogiovanni G, Bucci N, De Canio A, Indrio F, Cavallo L, Ierardi E, Miniello VL. Inhibition of Helicobacter pylori infection in humans by Lactobacillus reuteri ATCC 55730 and effect on eradication therapy: a pilot study. Helicobacter. 2008 Apr;13(2):127-34. doi: 10.1111/j.1523-5378.2008.00593.x. PMID 18321302